CLINICAL TRIAL: NCT05132439
Title: Metformin BenefIts Lower Extremities With Intermittent Claudication (MOBILE_IC)
Brief Title: MetfOrmin BenefIts Lower Extremities With Intermittent Claudication
Acronym: MOBILE IC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other); Northwestern University (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARB-012-20F; I01CX002150 (NIH)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Intermittent Claudication
Keywords: Peripheral artery disease; intermittent claudication; metformin; anti-inflammatory agents; clinical trial protocol; atherosclerosis
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease; Atherosclerosis | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Two arm randomization to 1000mg metformin ER or placebo daily with 1:1 parallel randomization, Randomization stratification will be based on baseline Maximum Walking Distance on the 6 Minute Walk Test and smoking status
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a triple-blinded randomized controlled trial. Therefore, the allocation of participants to either placebo or metformin is unknown by the participant, research personnel, and investigator. The study statistician will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin ER 1000mg (Experimental): daily by mouth
  Interventions: Drug: Metformin ER
- Matching placebo (Placebo Comparator): daily by mouth
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin ER — Oral medication typically used for Type 2 diabetes with presumed anti-inflammatory properties
  Other Names: Glucophage
  Arms: Metformin ER 1000mg
Drug: placebo — Matched to active study drug
  Arms: Matching placebo

SUMMARY:
Peripheral arterial disease (PAD) affects over 20% of aged adults and is very common among Veterans due significant tobacco use. PAD is due to the progressive blockage of peripheral arteries, predominantly to the legs, and results in intermittent claudication (IC) or recurrent muscle pain with activity secondary to insufficient blood supply. Those with PAD and IC experience a progressive decline in walking and poor quality of life. There is no effective medical treatment for PAD and IC. Metformin is a safe and effective treatment for Type 2 diabetes but it can also reduce inflammation, oxidative stress, and improve energy requirements as well as improve blood flow to the legs. Therefore, the investigators will test the ability of Metformin to improve overall functional status, reduce PAD progression, and reduce systemic inflammation in Veterans suffering from PAD and IC in a randomized, placebo controlled trial: Metformin BenefIts Lower Extremities with Intermittent Claudication (MOBILE IC) Trial. The success of this trial may identify a safe and effective treatment for PAD and IC.

DETAILED DESCRIPTION:
This is a quadruple blinded randomized controlled trial. Therefore, the allocation of participants to either placebo or metformin is unknown by the participant, research personnel, investigator, or blinded statistician. A total of 200 participants will be randomized over the course of 3 years. Study drug is administered to participants after all inclusion and no exclusion criteria is confirmed, informed consent is completed, and they are randomized. Study drug is continued throughout for 6 months following randomization. Participants are prospectively observed and monitored for 12 months after randomization. The patients' involvement (study visits/study phone calls) will last 12 months. Then, for 5 years, the study team will do a medical chart review as outlined in the ICF and protocol. All main study endpoints are within the 12-month time point. Secondary endpoints including MACE and MALE - major adverse cardiac and major adverse limb events - are time to event end points which can continue beyond the 12-month study time frame and will inform not only the effect of metformin on IC but also the natural history of IC among patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Veteran >35 & <89
* Symptoms of Intermittent claudication
* Medically stable, optimal medical therapy (for >3 months prior to randomization which includes - statin and anti-platelet therapy, blood pressure control, smoking cessation and physical activity counseling)

  a. Participants may not comply with the above measures to meet inclusion criteria, but investigator driven attempts to maximize the optimal medical therapy, as tolerated, for each participant prior to trial enrollment
* PAD as defined by ABI <0.9 or >0.9 with evidence of PAD as documented by pulse volume recordings (within 6 months prior to expected randomization date)
* Maximum Walking Distance (MWD) on the 6-minute walk test (6MWT) of greater than or equal to 50 meters with onset of pain before or at 400 meters without the use of a walker (cane is acceptable; within 6 months of expected randomization date)

Exclusion Criteria:

* Diabetes (Type I or II) or Hemoglobin A1c>6.5 (within 6 months of expected randomization)
* Currently Taking metformin or have previously taken metformin (within 6 months of enrollment)
* Medical condition that limit their ability to ambulate other than PAD (i.e., Angina, CHF, pulmonary disease requiring oxygen, malignancy requiring treatment, etc.)
* Prior above or below knee amputation
* Critical limb threatening ischemia (i.e., non-healing wounds or rest pain)
* Planned hospital admission, major operation, or lower extremity revascularization to be completed (within 12 months after expected randomization date)
* Prior major operation or lower extremity revascularization (within the 3 months before expected randomization)
* Unable to complete quality of life testing due to Non-English Speaking and/or Dementia
* Kidney disease - dialysis or eGFR<45 (within 6 months of expected randomization date)*
* Planned iodinated contrasted study (within 6 months of expected randomization date)
* Evidence current or history of hepatic failure
* Women who are pregnant or breast feeding
* Unable to swallow uncrushed pills
* Investigator expects inclusion could cause harm to subject

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximal Walking distance on the 6 minute walk test | 6 month
  This validated measure of functional status in PAD and IC is highly reproducible and the ideal measure of real-life walking capacity

SECONDARY OUTCOMES:
6 minute walk test | 6 month
  This validated measure of functional status in PAD and IC is highly reproducible and the ideal measure of real-life walking capacity. The six minute walk test includes maximal walking distance, pain free walking distance, time to pain onset.
6 minute walk test | 12 month
  This validated measure of functional status in PAD and IC is highly reproducible and the ideal measure of real-life walking capacity. The six minute walk test includes maximal walking distance, pain free walking distance, time to pain onset.
Cardiopulmonary exercise test | 6 month
  The CPET is a well validated, reproducible measure symptom-limited (maximal) aerobic and anaerobic capacity in patients with PAD and IC and correlates with systemic disease severity and outcome
Cardiopulmonary exercise test | 12 month
  The CPET is a well validated, reproducible measure symptom-limited (maximal) aerobic and anaerobic capacity in patients with PAD and IC and correlates with systemic disease severity and outcome
EndoPAT | 6 month
  Systemic endothelial cell function and health will be evaluated by EndoPAT, measuring peripheral artery tonometry and generates reproducible digital pulse wave amplitude before and during reactive hyperemia induced by brachial artery occlusion with a blood pressure cuff
Grip Strength | 6 month
  Grip strength with a dynamometer provides a digital reading of force
EndoPAT | 12 month
  Systemic endothelial cell function and health will be evaluated by EndoPAT, measuring peripheral artery tonometry and generates reproducible digital pulse wave amplitude before and during reactive hyperemia induced by brachial artery occlusion with a blood pressure cuff
Grip Strength | 12 month
  Grip strength with a dynamometer provides a digital reading of force
Ankle brachial index and pulse volume recording | 6 month
  The ABI and PVR assess regional lower extremity blood supply in large-vessels and contribution of collaterals
Ankle brachial index | 12 month
  The ABI assesses regional lower extremity blood supply in large-vessels and contribution of collaterals
Health related quality of life questionnaire | 6 month
  Functionality outcomes will be supported by the general (SF-36) and disease specific (Vascular Quality of Life Questionnaire [VascQol6]) health related quality of life questionnaires.
Health related quality of life questionnaires | 12 month
  Functionality outcomes will be supported by the general (SF-36) and disease specific (Vascular Quality of Life Questionnaire [VascQol6]) health related quality of life questionnaires.
Walking Impairment Questionnaire | 6 month
  A subjective measure of patient-reported walking performance developed for PAD
Walking Impairment Questionnaire | 12 month
  A subjective measure of patient-reported walking performance developed for PAD
Freedom from major cardiac and major limb events | 12 month
  Major cardiac events include: composite of CVD mortality, myocardial ischemia, coronary revascularization, hospitalization for heart failure, non-fatal stroke, and transient ischemic attack. Major adverse limb events include: composite of minor and major amputations, revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Edith I. Tzeng, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reitz KM, Althouse AD, Forman DE, Zuckerbraun BS, Vodovotz Y, Zamora R, Raffai RL, Hall DE, Tzeng E. MetfOrmin BenefIts Lower Extremities with Intermittent Claudication (MOBILE IC): randomized clinical trial protocol. BMC Cardiovasc Disord. 2023 Jan 21;23(1):38. doi: 10.1186/s12872-023-03047-8. PMID 36681798